CLINICAL TRIAL: NCT00434031
Title: Neoadjuvant Therapy With Trastuzumab and Docetaxel Followed by Trastuzumab, Caelyx (Liposomal Doxorubicin) and Cyclophosphamide in Operable or Locally Advanced Her-2 Positive Breast Cancer
Brief Title: CETRA: Neoadjuvant Caelyx and Trastuzumab in Her-2 Positive Breast Cancer
Acronym: CETRA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: National Cancer Institute, Naples (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CETRA; EudraCT number: 2006-003993-85
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: locally advanced; stage II; stage IIIa; stage IIIb; HER-2 positive; primary
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Trastuzumab; liposomal doxorubicin

INTERVENTIONS:
Drug: docetaxel
Drug: cyclophosphamide
Drug: trastuzumab
Drug: liposomal doxorubicin

SUMMARY:
The purpose of this study is to evaluate the rate of pathologic complete response when giving docetaxel and trastuzumab followed by caelyx (liposomal doxorubicin), cyclophosphamide and trastuzumab before surgery in treating women with operable or locally advanced HER-2 positive breast cancer.

DETAILED DESCRIPTION:
Chemotherapy in association with trastuzumab, a monoclonal antibody, given before surgery, has been shown to reduce tumor size and permit better resection of HER-2 positive breast cancers. This study will evaluate the activity of a neoadjuvant treatment with docetaxel and trastuzumab given every 3 weeks for 4 cycles, followed by the combination of caelyx, cyclophosphamide and trastuzumab every 3 weeks for 4 cycles. Patients will undergo breast cancer surgery 2-5 weeks after the completion of neoadjuvant therapy. Adjuvant therapy after surgery will be given according to existing guidelines, and will include an additional 10 cycles of trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast cancer
* Stage II-IIIB (T0-1-2-3-4-N+-M0 or T2-3-4-N0-M0; according to TNM AJCC classification, 2002)
* Hyperexpression of HER-2/neu (HercepTest 3+ or positive FISH test)
* Age> 18 e < 65 years
* Left ventricular ejection fraction (LVEF) > or = 55%
* ECOG Performance Status 0-2
* Neutrophils > or = 2000/mm³, platelets > or = 100.000/mm³ , hemoglobin > or = 10 g/dl), GOT, GPT and bilirubin < 1.25 x the upper normal limit, creatinine < 1.25 x the upper normal limit.
* Life expectancy > 3 months
* Signed informed consent.

Exclusion Criteria:

* Any prior treatment for breast cancer
* Metastatic disease (M1)
* Performance status (ECOG) > or = 3
* Current malignancy or history of prior malignancy within past 10 years (with the exception of adequately treated non-melanoma skin cancer and carcinoma in situ of the uterine cervix)
* Neutrophils < 2.000/mm³ , platelets < 100.000/mm³ , hemoglobin < 10 g/dl.
* Creatinine > 1.25 x the upper normal limit
* GOT and/or GPT and/or bilirubin >1.25 x the upper normal limit.
* Concomitant conditions that, in the investigator's opinion, contraindicate the use of the drugs in the protocol.
* Congestive heart failure or history of congestive heart failure, unstable angina pectoris, myocardial infarction, clinically significant valvulopathy or uncontrolled arrhythmias
* Active infection
* Incapacity or refusal to provide informed consent.
* Inability to comply with follow up
* Pregnant or nursing females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09

PRIMARY OUTCOMES:
complete pathologic response rate

SECONDARY OUTCOMES:
toxicity of neoadjuvant treatment
predictive ability of noninvasive diagnostic methods for results of neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Matteis, M.D., Principal Investigator — NCI Naples, Division of Medical Oncology C; Giuseppe D'Aiuto, M.D., Principal Investigator — NCI Naples, Division of Surgical Oncology A; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Unit
Locations (1):
- Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli, Italy